CLINICAL TRIAL: NCT01711814
Title: A Phase 2 Open-Label, Noncomparative, Multicenter Extension Study to Evaluate the Long-term Safety and Efficacy of ASP015K in Subjects Previously Enrolled in a Phase 2 ASP015K Rheumatoid Arthritis Study
Brief Title: A Study to Evaluate the Long-term Safety and Efficacy of ASP015K in Subjects Previously Enrolled in a Phase 2 ASP015K Rheumatoid Arthritis Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Astellas Pharma Global Development, Inc. (Industry)
Collaborators: Janssen Biotech, Inc. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 015K-CL-RA25; 2011-006021-23 (EudraCT Number)
Record Dates: First submitted 2012-10-19; First posted 2012-10-22 (Estimated); Last update posted 2024-10-21 (Actual); Status verified 2024-10

CONDITIONS: Arthritis, Rheumatoid
Keywords: Rheumatoid Arthritis; ASP015K
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — peficitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ASP015K (Experimental): Experimental
  Interventions: Drug: peficitinib

INTERVENTIONS:
Drug: peficitinib — oral
  Other Names: ASP015K

SUMMARY:
The purpose of this study is to evaluate the long-term safety and efficacy of ASP015K in subjects with Rheumatoid Arthritis (RA) who have completed a preceding Phase 2 ASP015K RA study.

DETAILED DESCRIPTION:
This study is comprised of a 104 week treatment period beginning on Day 1 of study drug administration and a 30-day follow-up period or permanent termination of clinical development of the product, whichever is earlier.

ELIGIBILITY:
Inclusion Criteria:

* Subject completed the week 12 visit in one of the Phase 2, ASP015K Rheumatoid Arthritis studies within the previous 14 days.
* Male and Female subjects must be willing to comply with contraception requirements as well as restrictions regarding egg and sperm donation

Exclusion Criteria:

* Subject has any condition considered by the Principal Investigator or Medical Monitor to preclude adequate evaluation of drug safety
* Subject is scheduled to receive any investigational drug other than ASP015K during the course of the study
* Subject is scheduled to receive a prohibited medication
* Subject has a planned major surgery
* Subject discontinued study drug due to meeting study drug discontinuation criteria prior to completion of the Week 12 visit in the preceding study or fulfills study drug discontinuation criteria at the final study visit of the preceding study
* Subject has out of range laboratory values within 14 days of the Day 1 study dosing
* Absolute lymphocyte count (ALC) < 500/mm3
* Creatine Phosphokinase (CPK) > 1.5 x upper limit of normal unless the level has been stable for at least 2 consecutive blood draws (at least 7 days apart), and subject does not have symptoms of muscle aching, weakness, or severe unusual muscle cramps

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 611 (Actual)
Dates: Start 2012-09-26 (Actual); Primary Completion 2016-03-25 (Actual); Study Completion 2016-03-25 (Actual)

PRIMARY OUTCOMES:
Safety assessed by recording of adverse events and clinical laboratory evaluations | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Senior Medical Director, Study Director — Astellas Pharma Global Development
Locations (51):
- United States (20):
  - Site US3218, Birmingham, Alabama
  - Site US828, La Jolla, California
  - Site US3227, Palm Desert, California
  - Site US219, Palo Alto, California
  - Site US3332, Santa Maria, California
  - Site US3331, Colorado Springs, Colorado
  - Site US1894, Jacksonville, Florida
  - Site US3232, Orlando, Florida
  - Site US702, Morton Grove, Illinois
  - Site US3226, Vernon Hills, Illinois
  - Site US3329, Elizabethtown, Kentucky
  - Site US291, Wheaton, Maryland
  - Site US3298, Hickory, North Carolina
  - Site US3300, Oklahoma City, Oklahoma
  - Site US345, Duncansville, Pennsylvania
  - Site US3304, Wyomissing, Pennsylvania
  - Site US3306, Knoxville, Tennessee
  - Site US3319, Austin, Texas
  - Site US3327, Chesapeake, Virginia
  - Site US3320, Clarksburg, West Virginia
- Belgium (2):
  - Site BE3387, Brussels
  - Site BE3314, Brussels
- Bulgaria (3):
  - Site BG3613, Burgas
  - Site BG3217, Plovdiv
  - Site BG3303, Sofia
- Colombia (5):
  - Site CO3326, Barranquilla, Atlantico
  - Site CO3297, Bogotá
  - Site CO2826, Bucamaranga
  - Site CO3450, Bucaramanga
  - Site CO3451, Cali
- Czechia (4):
  - Site CZ3388, Prague
  - Site CZ3376, Praha-Nusle
  - Site CZ3225, Uherské Hradiště
  - Site CZ3449, Zlín
- Hungary (6):
  - Site HU3461, Balatonfüred
  - Site HU3398, Békéscsaba
  - Site HU3302, Budapest
  - Site HU3448, Budapest
  - Site HU3462, Budapest
  - Site HU3447, Debrecen
- Mexico (4):
  - Site MX3238, Guadalajara
  - Site MX3307, Guadalajara, Jalisco
  - Site MX3310, México
  - Site MX3317, Morelia
- Poland (7):
  - Site PL3233, Bialystok, Polska
  - Site PL3391, Bialystok
  - Site PL2893, Bydgoszcz
  - Site PL3603, Krakow
  - Site PL3601, Lublin
  - Site PL3600, Warsaw
  - Site PL3599, Warsaw

IPD SHARING:
Plan to Share IPD: Yes
Access to anonymized individual participant level data collected during the study, in addition to study-related supporting documentation, is planned for studies conducted with approved product indications and formulations, as well as products terminated during development. Studies conducted with product indications or formulations that remain active in development are assessed after study completion to determine if Individual Participant Data can be shared. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Access to participant level data is offered to researchers after publication of the primary manuscript (if applicable) and is available as long as Astellas has legal authority to provide the data.
Access Criteria: Researchers must submit a proposal to conduct a scientifically relevant analysis of the study data. The research proposal is reviewed by an Independent Research Panel. If the proposal is approved, access to the study data is provided in a secure data sharing environment after receipt of a signed Data Sharing Agreement.
URL: https://www.clinicaltrials.astellas.com/transparency/

REFERENCES:
- [Derived] Genovese MC, Greenwald MW, Gutierrez-Urena SR, Cardiel MH, Poiley JE, Zubrzycka-Sienkiewicz A, Codding CE, Wang A, He W, Amos R, Vinueza R, Wang X, Garg JP, Kivitz AJ. Two-Year Safety and Effectiveness of Peficitinib in Moderate-To-Severe Rheumatoid Arthritis: A Phase IIb, Open-Label Extension Study. Rheumatol Ther. 2019 Dec;6(4):503-520. doi: 10.1007/s40744-019-00167-6. Epub 2019 Aug 13. PMID 31410787
- See also: Link to results on the Astellas Clinical Study Results website — https://astellasclinicalstudyresults.com/study.aspx?ID=324